CLINICAL TRIAL: NCT01181401
Title: Randomized Phase II Study of Two Different Regimens of TPF Induction Chemotherapy Regimen Followed by Radiation Therapy Plus Cetuximab (TPF-CET-HART) vs. HART and Cis-platinum, 5-FU (PF-HART) in Patients With Locally Advanced Unresectable Squamous Cell Carcinomas of the Head and Neck
Brief Title: InductionChemo-Radio-Antibody-Treatment
Acronym: ICRAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Carmen Stromberger, Prof. Dr. Volker Budach, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT No. 2010-019347-18
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Squamous Cell Carcinoma of the Head; Squamous Cell Carcinoma of the Neck
Keywords: induction chemotherapy; radiotherapy; locally advanced head neck tumor; toxicity; LA SCCHN; Unresectable squamous cell cancer of the head and neck,; Stage IV (UICC)
MeSH Terms: interventions — Docetaxel; Cisplatin; Cetuximab; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TPF standard (Active Comparator): TPF version 1 (standard)
  1. Induction chemotherapy:
     Docetaxel 75 mg/m2 d 1 Cis-platinum 75 mg/m2 d 1 5-FU 750 mg/m2/d c.i. d 1-4 every 21 days for 3 cycles
  2. Antibody therapy with:
     cetuximab loading dose of 400 mg/m2 1 week prior to RTX, and 250 mg/m2 weekly x 6 concurrent to RTX
  3. RTX: HART (72 Gy), IMRT or 3D-conformal techniques
  Interventions: Drug: TPF induction chemotherapy
- TPF experimental (Experimental): TPF version 2 (experimental)
  1. Induction chemotherapy:
     Docetaxel 40 mg/m2 d 1+8 Cis-platinum 40 mg/m2 d 1+8 5-FU 1500 mg/m2/24h c.i. d 1+8 every 21 day for 3 cycles
  2. Antibody therapy with:
     cetuximab loading dose of 400 mg/m2 1 week prior to RTX, and 250 mg/m2 weekly x 6 concurrent to RTX
  3. RTX: HART (72 Gy), IMRT or 3D-conformal techniques
  Interventions: Drug: TPF experimental
- Standard RCT (Active Comparator): Standard RCT:
  1. HART (72 Gy), IMRT or 3D-conformal techniques
  2. with concurrent chemotherapy: Cis-platinum 30 mg/m2 once weekly d 1, 8, 15, 22, 29, 36 5-FU 600mg/m² /24h c.i. d 1-5
  Interventions: Radiation: Standard Radiochemotherapy (HART)

INTERVENTIONS:
Drug: TPF induction chemotherapy — Docetaxel 75 mg/m2 d 1 Cis-platinum 75 mg/m2 d 1 5-FU 750 mg/m2/d c.i. d 1-4 Cetuximab loading dose of 400 mg/m2 1 week prior to RTX, and 250 mg/m2 weekly x 6 concurrent to RTX
  Other Names: Docetaxel (Taxotere); Cisplatin; 5-Flurouracil; Cetuximab (Erbitux)
  Arms: TPF standard
Drug: TPF experimental — Docetaxel 40 mg/m2 d 1+8 Cis-platinum 40 mg/m2 d 1+8 5-FU 1500 mg/m2/24h c.i. d 1+8 every 21 day for 3 cycles 2. Antibody therapy with: cetuximab loading dose of 400 mg/m2 1 week prior to RTX, and 250 mg/m2 weekly x 6 concurrent to RTX
  Other Names: Docetaxel (Taxotere); Cisplatin; 5-Flurouracil; Certuximab
  Arms: TPF experimental
Radiation: Standard Radiochemotherapy (HART) — Hyperfractionated accelerated radiotherapy with concurrent Cisplatin and 5-Fluorouracil chemotherapy
  Other Names: Cis-platinum; 5-FU
  Arms: Standard RCT

SUMMARY:
This is an open-label, randomized, Phase II-study to evaluate the efficacy of a standard-TPF induction chemotherapy (IC) and an alternative TPF induction chemotherapy followed by radio-antibody-therapy, in patients with unresectable LA-SCC of the HN region (oro-hypopharynx carcinoma, cancer of the oral cavity).

The primary objective of the study is to assess the feasibility of an experimental 'fractionated' TPF regimen compared to a current standard TPF regimen.

Composite endpoint of compliance and feasibility in terms of

* response (RECIST1.1) and
* hematological acute toxicity (CTCAE v.4.02)
* on time application of RAT following an experimental or standard TPF IC.

Secondary endpoints are

* Treatment intensity achieved
* Toxicity (according to CTCAE v.4.02)
* Response rates after completion of induction chemotherapy and after completion of entire protocol treatment (RECIST1.1)
* Survival (progression-free, metastasis-free, recurrence-free, overall) 1 year after randomisation
* Quality of life according to EORTC QoL C30 & HN35

The study will be conducted at 5-6 investigational sites in Germany recruiting 90 patients in total. Eligible patients will have a diagnosis of histologically confirmed SSC of the HN. Patients will receive one of 2 different regimens of TPF IC followed by cetuximab together with radiotherapy (RAT) or a standard radiochemotherapy(RCT) regimen.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven unresectable SCC of the oral cavity, oropharynx and hypopharynx (stage IVA & IVB)
* Written and signed informed consent
* Karnofsky PS > 70 %
* Age ≥ 18 years
* Curative treatment intent
* Adequate bone marrow, hepatic and renal functions as evidenced by the following:

Hematology (Bone marrow):

* Neutrophils > 2.0 109/L
* Platelets > 100 x 109/L
* Hemoglobin > 10 g/dL

Hepatic function:

* Total serum bilirubin < 1 time the UNL of the participating center
* ASAT (SGOT) and ALAT (SGPT) < 2.5 x UNL
* Alkaline phosphatase < 5 x UNL

Renal function :

* serum creatinine (SC) < 120 µmol/L (1.4 mg/dl);
* if values are > 120 µmol/L, the creatinine clearance should be > 60 ml/min (actual or calculated by the Cockcroft-Gault method as follows :

weight (kg) x (140 - age) --------------------------------- K x serum creatinine

serum creatinine in mg/dL: K = 72 in man K = 85 in woman serum creatinine in µmol/L: K = 0.814 in man K = 0.96 in woman

• If of childbearing potential, willingness to use effective contraceptive method for the study duration and 2 months post-dosing.

All patients require:

* dental examination and appropriate dental preservation if needed 1 week prior to the beginning of radiotherapy,
* gastric feeding tube and Portal-catheter.

Exclusion Criteria:

* Other neoplasia within the past 5 years with the exception of a controlled skin cancer or "in situ" cervix cancer
* Unknown primary (CUP), nasopharynx, laryngeal or salivary gland cancer
* Distant metastatic disease (M1)
* Serious co-morbidity, e.g. arteriosclerosis with apoplexy, recent myocardial infarction, high-grade carotid stenoses, unstable cardiac disease despite treatment, congestive heart failure NYHA grade 3 and 4, insulin-dependent diabetes mellitus, uncontrolled hypertension, liver cirrhosis (Quick < 75%, total protein <3.0 g/dl, bilirubin >2mg/ml) or kidney insufficiency (creatinine >1.4 mg/ml, the creatinine clearance should be > 60 ml/min)
* patients with ASAT or ALAT > 2.5 UNL associated with alkaline phosphatase > 5 UNL are not eligible for the study
* Known HIV-infection
* Pregnancy or lactation
* Women of child-bearing potential with unclear contraception
* Previous treatment of the disease with chemotherapy, radiotherapy, EGFR-targeting agents or surgery exceeding biopsy in head and neck
* Concurrent treatment with other experimental drugs or participation in another clinical trial with any investigational drug within 30 days prior to study screening
* Social situations that limit compliance with study requirements
* Deficient dental preservation status or not accomplished wound healing
* Legal incapacity
* Prior accommodation in an institution under officially or judicially orders (§ 40 1 p. 3 No. 4 AMG)
* Symptomatic peripheral neuropathy National Cancer Institute-Common Toxicity Criteria (NCI-CTC) grade 2 and/or ototoxicity grade 2, except if due to trauma or mechanical impairment due to tumor mass
* Known allergic/hypersensitivity reaction to any of the components of the treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2010-08; Primary Completion 2015-04 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Feasibility of an experimental 'fractionated' TPF regimen compared to a current standard TPF regimen. | August 2010- December 2012
  acute hematological toxicity

SECONDARY OUTCOMES:
Survival and late morbidity | 1 year
  All adequate items illustrating acute toxicity and late morbidity, in particular by hematological measures until one year after treatment (according to NCI-CTCAE v.4.02) Survival (progression-free, metastases-free, recurrence-free, Overall survival) after 1 year Response rates after TPF IC (RECIST1.1) Response rates after completion of multimodal treatment (see follow-up for scheduling RECIST1.1) Efficacy in relation to HPV status (p16 IHC) Quality of life according to EORTC QLC-30 & HN35

CONTACTS AND LOCATIONS:
Overall Officials: Volker Budach, MD, PhD, Principal Investigator — Charité Universitaetsmedizin Berlin
Locations (5):
- Germany (5):
  - Charité Universitaetsmedizin Berlin, CVK, CBF, Berlin
  - University Medical Center Hamburg - Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Gießen und Marburg, Marburg
  - Universitätsklinikum Regensburg, Regensburg

REFERENCES:
- [Result] Vermorken JB, Remenar E, van Herpen C, Gorlia T, Mesia R, Degardin M, Stewart JS, Jelic S, Betka J, Preiss JH, van den Weyngaert D, Awada A, Cupissol D, Kienzer HR, Rey A, Desaunois I, Bernier J, Lefebvre JL; EORTC 24971/TAX 323 Study Group. Cisplatin, fluorouracil, and docetaxel in unresectable head and neck cancer. N Engl J Med. 2007 Oct 25;357(17):1695-704. doi: 10.1056/NEJMoa071028. PMID 17960012
- [Result] Posner MR, Hershock DM, Blajman CR, Mickiewicz E, Winquist E, Gorbounova V, Tjulandin S, Shin DM, Cullen K, Ervin TJ, Murphy BA, Raez LE, Cohen RB, Spaulding M, Tishler RB, Roth B, Viroglio Rdel C, Venkatesan V, Romanov I, Agarwala S, Harter KW, Dugan M, Cmelak A, Markoe AM, Read PW, Steinbrenner L, Colevas AD, Norris CM Jr, Haddad RI; TAX 324 Study Group. Cisplatin and fluorouracil alone or with docetaxel in head and neck cancer. N Engl J Med. 2007 Oct 25;357(17):1705-15. doi: 10.1056/NEJMoa070956. PMID 17960013
- [Result] Haddad R, Colevas AD, Tishler R, Busse P, Goguen L, Sullivan C, Norris CM, Lake-Willcutt B, Case MA, Costello R, Posner M. Docetaxel, cisplatin, and 5-fluorouracil-based induction chemotherapy in patients with locally advanced squamous cell carcinoma of the head and neck: the Dana Farber Cancer Institute experience. Cancer. 2003 Jan 15;97(2):412-8. doi: 10.1002/cncr.11063. PMID 12518365
- [Result] Bonner JA, Harari PM, Giralt J, Cohen RB, Jones CU, Sur RK, Raben D, Baselga J, Spencer SA, Zhu J, Youssoufian H, Rowinsky EK, Ang KK. Radiotherapy plus cetuximab for locoregionally advanced head and neck cancer: 5-year survival data from a phase 3 randomised trial, and relation between cetuximab-induced rash and survival. Lancet Oncol. 2010 Jan;11(1):21-8. doi: 10.1016/S1470-2045(09)70311-0. Epub 2009 Nov 10. PMID 19897418